CLINICAL TRIAL: NCT00356187
Title: Beta-blockade Reduces Catabolism in Severely Injured Trauma Patients
Brief Title: Beta Blockade in Critical Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment, end of funding
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03 DK73349 (completed); R03DK073349 (NIH)
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Propranolol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Propranol Treatment (Experimental)
  Interventions: Drug: Propranolol
- Standard of Care (No Intervention)

INTERVENTIONS:
Drug: Propranolol
  Arms: Propranol Treatment

SUMMARY:
Critically injured patients endure a period of hypermetabolism/catabolism after being resuscitated. The metabolic cost of this may be measured in loss of lean body mass, poor wound healing, susceptibility to infection and long hospital stays. While there have been some data to suggest that hypermetabolism can be ameliorated in burn patients by beta blockade, to our knowledge, a prospective trial in trauma patients has not yet been done. Our hypothesis is that nonselective beta blockade will reduce catabolism, improve glucose control, blunt loss of lean body mass, decrease infections and improve outcome in a cohort of critically injured patients.

ELIGIBILITY:
Inclusion Criteria:

* ISS>25, stable at 48 hours after injury
* Fully resuscitated
* Ventilated

Exclusion Criteria Include:

* Intracranial hypertension requiring active treatment
* Hypotension/Pressors
* Already on beta blocker for a standard indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-02-15 (Actual); Primary Completion 2009-01-31 (Actual); Study Completion 2009-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Insufficient enrollment to derive any results. Study closed in 2009 and is past data retention.
Groups:
- Propranol Treatment: Propranolol
- Standard of Care: Results: 0
  Insufficient enrollment to derive any results. Study closed in 2009 and is past data retention. PI has left institution and does not have any access to any data.
Period: Overall Study
Arm/Group | Propranol Treatment | Standard of Care
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Insufficient enrollment to derive any results. Study closed in 2009 and is past the HIPAA data retention date. PI has left institution and does not have any access to any data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranol Treatment | Standard of Care | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in REE vs. Controls
Time Frame: ICU admission date to ICU discharge or death
Population: Insufficient enrollment to derive any results. Study closed in 2009 and is past data retention. PI has left institution and does not have any access to any data.
Arm/Group | Propranol Treatment | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Changes in Protein Metabolism Measurements
Description: net nitrogen balance, fat-free mass, and fat mass
Time Frame: ICU admission date to ICU discharge or death
Population: as for outcome 1
Arm/Group | Propranol Treatment | Standard of Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Alterations in Neuroendocrine and Immunoinflammatory Measurements
Description: blood glucose levels, insulin requirements, cortisol levels, IL-6 and IL-10 levels, infection rates, and organ dysfunction
Time Frame: ICU admission date to ICU discharge or death
Population: as for outcome 1
Arm/Group | Propranol Treatment | Standard of Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Clinical Outcome Measurements
Description: Ventilator days, ICU and hospital days, and in-hospital mortality
Time Frame: ICU admission date to ICU discharge or death
Population: as for outcome 1
Arm/Group | Propranol Treatment | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Insufficient enrollment to derive any results. Study closed in 2009 and is past the HIPAA data retention date. PI has left institution and does not have any access to any data.
Arm/Group | Propranol Treatment | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No